CLINICAL TRIAL: NCT02556268
Title: Potential Pharmacokinetic Interaction of Human Immunodeficiency Virus (HIV) Antiretroviral Agents as Fixed-dose Combinations and Riociguat in HIV Patients
Brief Title: Interaction With HIV Antiretroviral Agents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17957
Record Dates: First submitted 2015-09-21; First posted 2015-09-22 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: HIV-DDI
Keywords: Single-Dose, Open-Label, Non-Blinded, Non-Placebo-; Controlled, Stratified Design
MeSH Terms: interventions — riociguat; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine, Rilpivirine, Tenofovir Drug Combination; Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; abacavir, dolutegravir, and lamivudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Riociguat and ATRIPLA (Experimental)
  Interventions: Drug: Riociguat (Adempas, BAY 63-2521); Drug: ATRIPLA
- Riociguat and COMPLERA (Experimental)
  Interventions: Drug: Riociguat (Adempas, BAY 63-2521); Drug: COMPLERA
- Riociguat and STRIBILD (Experimental)
  Interventions: Drug: Riociguat (Adempas, BAY 63-2521); Drug: STRIBILD
- Riociguat and TRIUMEQ (Experimental)
  Interventions: Drug: Riociguat (Adempas, BAY 63-2521); Drug: TRIUMEQ
- Riociguat and antiretroviral protease inhibitor with TRIUMEQ (Experimental)
  Interventions: Drug: Riociguat (Adempas, BAY 63-2521); Drug: Antiretroviral protease inhibitor

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY 63-2521) — 0.5 mg, Oral (fasted conditions), 1 single dose
Drug: ATRIPLA — 600 mg efavirenz, 200 mg emtricitabine, and 300 mg tenofovir disoproxil fumarate, i.e. 1 tablet, once daily
  Arms: Riociguat and ATRIPLA
Drug: COMPLERA — 200 mg emtricitabine, 25 mg rilpivirine, and 300 mg tenofovir disoproxil fumarate, i.e. 1 tablet, once daily
  Arms: Riociguat and COMPLERA
Drug: STRIBILD — 150 mg elvitegravir, 150 mg cobicistat, 200 mg emtricitabine, and 300 mg tenofovir disoproxil fumarate, i.e. 1 tablet, once daily
  Arms: Riociguat and STRIBILD
Drug: TRIUMEQ — 600 mg abacavir, 50 mg dolutegravir, and 300 mg lamivudine, i.e. 1 tablet, once daily
  Arms: Riociguat and TRIUMEQ
Drug: Antiretroviral protease inhibitor — Any approved antiretroviral protease inhibitor such as atazanavir, darunavir, indinavir, ritonavir, and saquinavir ; consistent with the most recent prescribing information documents
  Arms: Riociguat and antiretroviral protease inhibitor with TRIUMEQ

SUMMARY:
To investigate the pharmacokinetic drug-drug interaction potential of fixed dose antiretroviral therapies, i.e. ATRIPLA, COMPLERA, STRIBILD, TRIUMEQ, or any approved antiretroviral protease inhibitor in combination with (preferably) TRIUMEQ, on the exposure to riociguat in HIV patients on a stable dose of one of these therapies.

• To Assess the safety and tolerability of riociguat treatment in combination with these fixed-dose antiretroviral therapies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged >=18 to <65 years with a confirmed diagnosis of HIV receiving a stable regimen of ATRIPLA, COMPLERA, STRIBILD, TRIUMEQ, or any approved antiretroviral protease inhibitor such as atazanavir, darunavir, indinavir, ritonavir, and saquinavir in combination with (preferably) TRIUMEQ consistent with the most recent prescribing information documents for at least 6 weeks before concomitant administration of a single oral dose of 0.5 mg riociguat
* No clinical evidence of pulmonary hypertension
* Written informed consent

Exclusion Criteria:

* Severe diseases for which it can be assumed that the pharmacokinetics or effects of the study drug will not be normal
* History of coronary artery disease
* Symptomatic postural hypotension (e.g. dizziness, lightheadedness)
* History of bronchial asthma or any other airway disease
* Renal impairment with creatinine clearance <15 mL/min
* Severe hepatic impairment (Child-Pugh class C)
* Systolic blood pressure below 100 mmHg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02-23 (Actual); Primary Completion 2016-12-07 (Actual); Study Completion 2016-12-07 (Actual)

PRIMARY OUTCOMES:
AUC of riociguat | at pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8 24 and 48 hours post-dose
Cmax of riociguat | at pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8 24 and 48 hours post-dose
AUC of riociguat main metabolite M1 (BAY 60-4552) | at pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8 24 and 48 hours post-dose
Cmax of riociguat main metabolite M1 (BAY 60-4552) | at pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8 24 and 48 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- United States (2):
  - Orlando, Florida
  - Boston, Massachusetts